CLINICAL TRIAL: NCT06065904
Title: Exploring the Efficacy of a Comprehensive Nutritional Intervention for Children With Cerebral Palsy and ASD: A Randomized Controlled Trial at a Single Center
Brief Title: Randomized One-Center Controlled Trial on a Comprehensive Nutritional Intervention for Children With Cerebral Palsy and ASD
Acronym: Nutrilect
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Silviya Pavlova Nikolova, PhD (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor-Investigator, Silviya Pavlova Nikolova, PhD, The research is financed by the European Union-NextGenerationEU, through the National Recovery and Resilience Plan of the Republic of Bulgaria, project № BG-RRP-2.004-0009-C02., Medical University of Varna
Organization: Medical University of Varna (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: MUVarna
Record Dates: First submitted 2023-09-16; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Nutrition Disorder, Child
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CP with recommended diet (Experimental): CP children that will follow a recommended menu
  Interventions: Behavioral: Nutrilect
- CP with a standard of care nutritional menu (No Intervention): Children with CP that will not be advised on a specific menu
- ASD with recommended diet (Experimental): Children with ASD that will not be advised on a specific menu
  Interventions: Behavioral: Nutrilect
- ASD with a standard of care nutritional menu (No Intervention): Children with ASD that will not be advised on a specific menu

INTERVENTIONS:
Behavioral: Nutrilect — This intervention involves a comprehensive approach that includes a thorough nutritional assessment and individualized nutrition plan for children with cerebral palsy (CP) and Autism Spectrum Disorder (ASD), addressing their unique dietary needs and challenges. It encompasses nutritional counseling, dietary modifications when necessary, and seamless integration with other therapies, including speech therapy and psychological consultation. The overarching goal is to optimize growth, muscle function, and overall well-being in these children by providing tailored nutritional support alongside a holistic care approach.
  Arms: ASD with recommended diet; CP with recommended diet

SUMMARY:
The study is a prospective, single-center, randomized controlled trial that will be conducted at the Medical University of Varna. This setting offers access to a wealth of clinical expertise in managing CP and ASD and a rich tradition of conducting robust nutritional interventions.

ELIGIBILITY:
Inclusion Criteria:

* A formal diagnosis made by a qualified neurologist. The diagnosis can span across the different types of CP and ASD.
* Expressed willingness to participate in the study.
* Availability for the entire duration of the study.

Exclusion Criteria:

* Children with acute medical conditions or comorbidities that may significantly disrupt study assessments.
* Any severe infections within the last 10 days prior to the study.
* Presence of genetic syndromes that could influence nutritional status, e.g., Silver Russel syndrome or Down syndrome.
* Parents with cognitive impairments, which might pose challenges in their participation during assessments/intervention.
* Children who have been part of any major dietary or nutritional interventions in the last three months.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-12-23 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
bedridden days monthsmean duration of bedridden days over six months | six months
  mean duration of bedridden days

SECONDARY OUTCOMES:
Weight-for-Age Z-Score | six months
  The Weight-for-Age Z-Score serves as a secondary outcome measure in the study, primarily focusing on assessing changes in the study participants' weight status. Data collection involves anthropometric assessments and the utilization of reference growth charts, specifically the World Health Organization (WHO) reference charts, to record participants' weight relative to their age. This measurement employs the Z-score as the unit of measure, quantifying deviations in weight from the baseline. A positive Z-score indicates above-average weight for a given age group, while a negative Z-score indicates below-average weight, providing a valuable indicator of participants' nutritional status and growth trends over time.
Height-for-Age Z-Score | six months
  The Height-for-Age Z-Score is a secondary outcome measure focused on evaluating changes in the study participants' height status. It involves anthropometric assessments and the use of WHO reference growth charts to record participants' height in relation to their age. The Z-score is the unit of measure, allowing for the quantification of height changes relative to the baseline. A positive Z-score indicates above-average height for the age group, while a negative Z-score indicates below-average height, offering a valuable indicator of participants' growth patterns and nutritional well-being over time.
BMI-for-Age Z-Score | six months
  The secondary outcome measure, BMI-for-age Z-Score, assesses changes in the study participants' Body Mass Index (BMI) in relation to their age. This measurement relies on deriving BMI from weight and height measurements, with comparisons made using reference growth charts provided by the World Health Organization (WHO). The Z-score is employed as the unit of measure, enabling the quantification of BMI changes relative to the baseline. A positive Z-score signifies an above-average BMI for the age group, whereas a negative Z-score indicates a below-average BMI, serving as an essential metric for tracking variations in participants' nutritional status and body composition throughout the study.
Number of social interactions per week with non-family members | six months
  The 'Number of Social Interactions per Week with Non-Family Members' is a quantitative measure that assesses the child's weekly engagement in social interactions with individuals outside their immediate family circle. It involves tracking and recording the frequency of diverse social exchanges, such as conversations, playdates, school-related interactions, and community engagements over a one-week period. This measure is instrumental in evaluating the child's social participation, integration into broader social networks, and overall quality of life. A higher number of interactions typically indicates greater social engagement and integration, while a lower number may signal reduced social participation, highlighting areas that require attention for the child's holistic development.
Total Number of New Spoken Words per Month | six months
  Total Number of New Spoken Words per Month is a quantitative measure employed to evaluate a child's language development and communication skills over a one-month period. This measure involves systematically counting and recording the distinct words that the child effectively uses and articulates in conversations, interactions, or observations during the course of each month. Specifically, it focuses on identifying and tallying newly acquired words within the given timeframe.A higher number of newly spoken words typically indicates positive language development, reflecting effective vocabulary expansion and improved communication skills. A threshold of one new word per month is established as a meaningful indicator of progress.
Total Days of School or Kindergarten Attendance per month | six month
  Total Days of School or Kindergarten Attendance per Month is a quantitative measure used to precisely assess a child's consistent participation in a formal educational setting, such as school or kindergarten, within the span of one month.A higher total number of days attended per month reflects more consistent participation in educational settings, indicating a stronger connection to learning opportunities and educational routines. Conversely, a lower total may indicate irregular attendance or potential challenges that require attention.
Number of Leisure Activities per Month | six months
  The 'Number of Leisure Activities per Month' is a quantitative measure used to assess children's level of engagement in leisure and recreational pursuits over a one-month period. This measure involves systematically counting and documenting the quantity of diverse leisure activities, hobbies, or pastimes that the individual participates in during the designated month. Leisure activities encompass a wide range of choices, such as hobbies, sports, cultural events, or entertainment, selected for relaxation, enjoyment, and personal enrichment. A higher count of leisure activities often indicates a more diversified and active leisure lifestyle, potentially contributing to an enhanced overall quality of life, while a lower count may suggest limited engagement in leisure pursuits, highlighting opportunities for greater leisure satisfaction.

IPD SHARING:
Plan to Share IPD: No